CLINICAL TRIAL: NCT01258348
Title: A Phase 1b Study of LY573636-sodium in Combination With Sunitinib Malate in Patients With Metastatic Renal Cell Cancer
Brief Title: A Phase 1b Trial in Patients With Renal Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10407; H8K-MC-JZAI (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY573636 +sunitinib (Experimental)
  Interventions: Drug: Drug: LY573636-sodium; Drug: Sunitinib

INTERVENTIONS:
Drug: Drug: LY573636-sodium — Participant specific dose based on height, weight and gender to target a specific exposure range, administered intravenously on Day 4 of a 42-day (6-week) cycle.
  Dose will be escalated to reach the maximum tolerated dose (MTD). A cohort of participants enrolled after MTD will receive albumin-tailored doses.
  Participants may continue on treatment until clinical or objective disease progression.
  Other Names: Tasisulam
Drug: Sunitinib — 37.5 or 50 milligrams (mg), administered orally, daily for a 42-day (6-week) cycle.
  Participants may continue on treatment until clinical or objective disease progression.

SUMMARY:
The purpose of this study is to determine a safe dose of LY573636-sodium to be given in combination with sunitinib to patients with metastatic Renal Cell Carcinoma (RCC) and to determine any side effects that may be associated with LY573636-sodium and sunitinib combination in this patient population. The tumor response rate will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed diagnosis of metastatic Renal Cell Carcinoma (RCC)
* Participants must have received no prior treatment with a cytotoxic-based chemotherapy regimen
* Participants must have measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines
* Have adequate hematologic, hepatic and renal function
* Have a serum albumin level greater than equal to 3.0 grams/Liter (g/L)
* Participants with reproductive potential should use medically approved contraceptive precautions during the trial and for 6 months following the last dose of study drug
* Exhibit participant compliance and geographic proximity that allow for adequate follow-up
* Have given written informed consent approved by Lilly and the ethical review board (ERB)/institutional review board (IRB) governing the site
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy, for at least 4 weeks (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy (except alopecia). Participants who have received whole-brain radiation must wait 90 days before starting study therapy

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have received a prior cytotoxic chemotherapy-based systemic therapy for metastatic RCC
* Have had any of the following within 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure (CHF), cerebrovascular accident, transient ischemic attack, or pulmonary embolism
* Ongoing cardiac arrhythmias greater than New York Health Association Class II (Protocol Attachment JZAI.4), atrial fibrillation of any grade, or prolongation of the QTc interval to greater than 450 milliseconds (msec) for males or greater than 470 msec for females
* Have uncontrolled hypertension [greater than 150/100 millimeters of mercury (mm Hg) despite optimal medical therapy], or history of poor compliance with antihypertensive treatment
* Participants with documented central nervous system or leptomeningeal metastasis (brain metastasis) at the time of study entry. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before study entry
* Participants with serious concomitant OR pre-existing disorders, including active bacterial, fungal, or viral infection, incompatible with the study (at the discretion of the investigator)
* Participants receiving warfarin therapy for treatment of venous thrombosis or other prothrombotic conditions
* Participants with a second primary malignancy that could affect interpretation of the results. NOTE: Participants with adequately treated carcinoma of the skin (excluding melanoma) and participants with a prior history of malignancy who have been disease-free for greater than 2 years are eligible
* Participants who have previously completed or withdrawn from this study or any other study investigating LY573636
* Participants who have previously received sunitinib
* Participants who are unable to swallow capsules
* Participants who require concomitant use of potent Cytochrome P450 3A4 (CYP3A4) inducers or inhibitors
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon -Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the Participant Flow are the reasons the participant discontinued treatment. All participants who received at least 1 dose of study drug were considered to have completed the study.
Groups:
- LY 340 μg/mL + Sunitinib 50 mg: LY573636 to target a maximum concentration (Cmax) of 340 micrograms per milliliter (μg/mL) (LY 340 μg/mL) as a 2-hour infusion on Days 4 and 25 of a 6-week cycle and sunitinib 50 milligrams (mg) orally, daily for 4 weeks followed by 2 weeks with no sunitinib dosing.
- LY 300 μg/mL + Sunitinib 50/37.5 mg: LY573636 to target a Cmax of 300 μg/mL (LY 300 μg/mL) as a 2-hour infusion on Days 4 and 25 of a 6-week cycle and either sunitinib 50 mg orally, daily for 4 weeks followed by 2 weeks with no sunitinib dosing or sunitinib 37.5 mg daily continuously for 6 weeks .
- LY 320 μg/mL + Sunitinib 37.5 mg: LY573636 to target a Cmax of 320 μg/mL (LY 320 μg/mL) as a 2-hour infusion on Day 4 of a 6-week cycle and sunitinib 37.5 mg orally, daily continuously for 6 weeks.
- LY 340 μg/mL + Sunitinib 37.5 mg: LY573636 to target a Cmax of 340 μg/mL (LY 340 μg/mL) as a 2-hour infusion on Day 4 of a 6-week cycle and sunitinib 37.5 mg orally, daily continuously for 6 weeks.
- LY 360 μg/mL + Sunitinib 37.5 mg: LY573636 to target a Cmax of 360 μg/mL (LY 360 μg/mL) as a 2-hour infusion on Day 4 of a 6-week cycle and sunitinib 37.5 mg orally, daily continuously for 6 weeks.
Period: Overall Study
Arm/Group | LY 340 μg/mL + Sunitinib 50 mg | LY 300 μg/mL + Sunitinib 50/37.5 mg | LY 320 μg/mL + Sunitinib 37.5 mg | LY 340 μg/mL + Sunitinib 37.5 mg | LY 360 μg/mL + Sunitinib 37.5 mg
Started | 1 | 5 | 3 | 6 | 6
Received at Least 1 Dose of Study Drug | 1 | 5 | 3 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 5 | 3 | 6 | 6
Not completed — Adverse Event | 1 | 1 | 3 | 2 | 4
Not completed — Progressive Disease | 0 | 3 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: LY573636 dose was to target a specific maximum concentration (Cmax) as a 2-hour infusion on Days 4 and 25 or Day 4 of a 6-week cycle. Sunitinib 50 milligrams (mg) orally, daily for 4 weeks followed by 2 weeks with no sunitinib dosing or sunitinib 37.5 mg daily continuously for 6 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 61.4 [40.4 to 75.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African | 2
  Race: Caucasian | 17
  Race: East Asian | 1
  Race: Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose for Phase 2 Studies of LY573636-Sodium Combined With Sunitinib in Participants With Metastatic Renal Cell Carcinoma
Description: Recommended Phase 2 dose was determined by maximum tolerated dose (MTD). MTD is the highest dose with <33% of participants having a dose-limiting toxicity (DLT) during the first 6-week cycle of treatment. DLT is an adverse event (AE) that is likely related to study drug or combination and fulfills any 1 of the following: Common Terminology Criteria for AE (CTCAE, Version 3.0) Grade (Gr) 4 neutropenia lasting ≥5 days; Gr 4 neutropenia with fever; Gr 4 thrombocytopenia; Gr ≥3 thrombocytopenia with bleeding; Gr ≥3 nonhematologic toxicity (excluding controllable nausea/vomiting or diarrhea and alopecia); Gr 3 electrolyte toxicity that is not resolved with standard treatments; Gr ≥3 elevated hepatic enzyme abnormalities in the setting of preexisting hepatic metastasis may not be considered a DLT; a DLT can be declared if a participant experiences increasing toxicity during treatment.
Time Frame: Predose up to 42 days postdose in Cycle 1 (6 weeks per cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: micrograms per milliliter (μg/mL)
Arm/Group | LY 340 μg/mL + Sunitinib 50 mg | LY 300 μg/mL + Sunitinib 50/37.5 mg | LY 320 μg/mL + Sunitinib 37.5 mg | LY 340 μg/mL + Sunitinib 37.5 mg | LY 360 μg/mL + Sunitinib 37.5 mg
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 6
micrograms per milliliter (μg/mL) | NA — MTD was not reached because the enrollment was stopped early. | NA — MTD was not reached because the enrollment was stopped early. | NA — MTD was not reached because the enrollment was stopped early. | NA — MTD was not reached because the enrollment was stopped early. | NA — MTD was not reached because the enrollment was stopped early.

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY573636
Description: Time frame: Cycle 1:day 4: pre-dose, start of infusion, end of infusion,30min,1h,2h,4h,6h,8h,10h,22h,46h,70h,166h,360h post infusion, day 25: predose, during infusion, end of infusion,30min,30min,1h,2h,4h,6h,8h,10h,22h,46h,70h,166h,360h post infusion.
Time Frame: Predose up to 2 hours postdose in Cycles 1 and 2 (6 weeks per cycle)
Population: Participants who received study drug and had sufficient pharmacokinetic (PK) data to estimate Cmax at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- LY573636: LY573636 dose was to target a specific maximum concentration (Cmax) as a 2-hour infusion on Days 4 and 25 or Day 4 of a 6-week cycle. Sunitinib 50 milligrams (mg) orally, daily for 4 weeks followed by 2 weeks with no sunitinib dosing or sunitinib 37.5 mg daily continuously for 6 weeks.
Arm/Group | LY573636
Number analyzed (Participants) | 21
micrograms per milliliter (µg/mL)
  Cycle 1 | 343.9 (10.7)
  Cycle 2: number analyzed (Participants) | 17
  Cycle 2 | 341.3 (16.1)

3. Secondary Outcome: Number of Participants With Tumor Responses
Description: Tumor response was assessed by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. Number of participants with tumor responses = number of participants with complete response (CR) + number of participants with partial response (PR). CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to end of treatment up to 66 weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY 340 μg/mL + Sunitinib 50 mg | LY 300 μg/mL + Sunitinib 50/37.5 mg | LY 320 μg/mL + Sunitinib 37.5 mg | LY 340 μg/mL + Sunitinib 37.5 mg | LY 360 μg/mL + Sunitinib 37.5 mg
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 6
Participants | 0 | 1 | 1 | 2 | 0

4. Secondary Outcome: Sunitinib Pharmacokinetics in the Presence of LY573636: Area Under the Curve (AUC)
Description: Time frame: Cycle 1 day 4: pre-dose, start of infusion, end of infusion,30min,1h,2h,4h,6h,8h,10h,22h,46h,70h,166h,360h post infusion, day 25: predose, during infusion, end of infusion,30min,30min,1h,2h,4h,6h,8h,10h,22h,46h,70h,166h,360h post infusion.
Time Frame: Days 1 to 42 in Cycle 1 (6 weeks per cycle)
Population: Participants who received sunitinib and had sufficient pharmacokinetic (PK) data to calculate AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (h*ng/mL)
Groups:
- Sunitinib: LY573636 dose was to target a specific maximum concentration (Cmax) as a 2-hour infusion on Days 4 and 25 or Day 4 of a 6-week cycle. Sunitinib 50 milligrams (mg) orally, daily for 4 weeks followed by 2 weeks with no sunitinib dosing or sunitinib 37.5 mg daily continuously for 6 weeks.
Arm/Group | Sunitinib
Number analyzed (Participants) | 13
hour*nanograms per milliliter (h*ng/mL) | 780.0 (51.1)

5. Secondary Outcome: Pharmacokinetics: Area Under the Curve of LY573636 Above the Albumin Corrected Threshold (AUCalb)
Description: LY573636 has been found to be highly bound to albumin. AUCalb is a surrogate measure of exposure to unbound (free) LY573636.
  Time frame: Cycle 1:day 4: pre-dose, start of infusion, end of infusion,30min,1h,2h,4h,6h,8h,10h,22h,46h,70h,166h,360h post infusion, day 25: predose, during infusion, end of infusion,30min,30min,1h,2h,4h,6h,8h,10h,22h,46h,70h,166h,360h post infusion.
  Cycle 2: predose and end of infusion.
Time Frame: Days 1 to 42 in Cycles 1 and Cycle 2 (6 weeks per cycle)
Population: Participants who received study drug and had sufficient pharmacokinetic (PK) data to calculate AUCalb at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter (h*µg/mL)
Arm/Group | LY573636
Number analyzed (Participants) | 21
hour*micrograms per milliliter (h*µg/mL)
  Cycle 1 | 241.3 (96.4)
  Cycle 2: number analyzed (Participants) | 17
  Cycle 2 | 866.3 (437.8)

6. Secondary Outcome: The Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and other non-serious adverse events. A summary of serious and all other non-serious adverse events is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion up to 70 weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY 340 μg/mL + Sunitinib 50 mg | LY 300 μg/mL + Sunitinib 50/37.5 mg | LY 320 μg/mL + Sunitinib 37.5 mg | LY 340 μg/mL + Sunitinib 37.5 mg | LY 360 μg/mL + Sunitinib 37.5 mg
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 6
Participants
  Serious Adverse Events | 1 | 2 | 2 | 3 | 1
  Other Nonserious Adverse Events | 1 | 5 | 3 | 6 | 6

ADVERSE EVENTS:
Arm/Group | LY 340 μg/mL + Sunitinib 50 mg | LY 300 μg/mL + Sunitinib 50/37.5 mg | LY 320 μg/mL + Sunitinib 37.5 mg | LY 340 μg/mL + Sunitinib 37.5 mg | LY 360 μg/mL + Sunitinib 37.5 mg
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/5 | 2/3 | 3/6 | 1/6
Other Adverse Events (participants affected / at risk) | 1/1 | 5/5 | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 340 μg/mL + Sunitinib 50 mg (N=1) | LY 300 μg/mL + Sunitinib 50/37.5 mg (N=5) | LY 320 μg/mL + Sunitinib 37.5 mg (N=3) | LY 340 μg/mL + Sunitinib 37.5 mg (N=6) | LY 360 μg/mL + Sunitinib 37.5 mg (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Appendicitis perforated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 340 μg/mL + Sunitinib 50 mg (N=1) | LY 300 μg/mL + Sunitinib 50/37.5 mg (N=5) | LY 320 μg/mL + Sunitinib 37.5 mg (N=3) | LY 340 μg/mL + Sunitinib 37.5 mg (N=6) | LY 360 μg/mL + Sunitinib 37.5 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 2 (3) | 2 (3) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 1 (1) | 2 (7) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 4 (6) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 4 (5) | 4 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 2 (4)
Asthenia (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 2 (2) | 5 (6) | 4 (4)
Infusion site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine colour abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 1 (1) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The primary outcome measure in this trial was not reached because the enrollment was stopped early before the maximum tolerated dose was reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days